CLINICAL TRIAL: NCT03569280
Title: A First-in-Human Study to Determine the Safety, Pharmacokinetics and Efficacy of KPG-121 When Administered With Enzalutamide, Abiraterone, or Apalutamide in Subjects With Non-Metastatic or Metastatic Castration-Resistant Prostate Cancer
Brief Title: Evaluation of Safety and Efficacy of KPG-121 Plus Enzalutamide, Abiraterone or Apalutamide in CRPC Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kangpu Biopharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KPG-121-101
Record Dates: First submitted 2018-05-22; First posted 2018-06-26 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Castration-Resistant Prostate Cancer
Keywords: KPG-121; Enzalutamide; Abiraterone; Apalutamide; Non-metastatic and Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; abiraterone

STUDY DESIGN:
Intervention Model Description: KPG-121 Plus Enzalutamide or Abiraterone or Apalutamid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- KPG-121 (Experimental): Safety and Antitumor Activity of KPG-121 capsules at different dose level for 21 days
  Interventions: Combination Product: Enzalutamide or Abiraterone or Apalutamid

INTERVENTIONS:
Combination Product: Enzalutamide or Abiraterone or Apalutamid — Antitumor treatment

SUMMARY:
This is a Phase 1, open-label, multicenter study of KPG-121 administered orally once daily (QD) in 28-day treatment cycles to adult subjects.

DETAILED DESCRIPTION:
This Phase 1 study will comprise two parts: Part 1 will be a 3+3 dose escalation design to characterize the MTD and a RP2D, Part 2 will be an expansion cohort at RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent provided prior to any study-related procedure being performed;
2. Able to swallow and retain orally administered medication;
3. Male aged 18 years and older;
4. diagnosis of prostate carcinoma;
5. Men with either non-metastatic or metastatic CRPC are eligible;
6. Completed at least 4 or more weeks of prior continuous therapy with fixed stable dose enzalutamide, abiraterone or apalutamide prior to initiating study treatment (for Part 1), or with fixed stable dose enzalutamide (for Part 2), with no change in dose for at least 2 weeks prior to screening;
7. Serum testosterone level <50 ng/dL (<0.5 ng/mL, <7.0 nmol/L).
8. ECOG performance status of 0 or 1;
9. Adequate baseline organ function;
10. Must have a QT interval corrected for heart rate according to Fridericia's formula (QTcF) <470 milliseconds (msec) or <480 msec with bundle branch block;
11. Male subject with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from time of screening until 3 months after the last dose of study medication;
12. Willing and able to comply with all protocol required visits and assessments.

Exclusion Criteria:

1. Prior chemotherapy, radiation;
2. Prior malignancy other than CRPC.
3. Uncontrolled hypothyroidism, or TSH >2.0 x ULN at screening.
4. Current use of or anticipated requirement of prohibited medication(s);
5. Any unresolved ≥grade 2 (per CTCAE v5.0) toxicity from previous anti-cancer therapy;
6. Previous history of difficulty swallowing capsules;
7. Known active infection requiring intravenous (IV);
8. Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test ;
9. History of seizure or any condition that may predispose subject to seizure (e.g., prior cortical stroke or significant brain trauma). History of loss of consciousness or transient ischemic attack within 12 months prior to the start of study medication;
10. Poorly controlled hypertension;
11. Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs
12. History or evidence of cardiovascular risk; known cardiac metastases;
13. Previous major surgery within 30 days prior to the start of study medication;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of KPG-121 | Cycle-1 (28-day)
  MTD is one dose level below the dose level that results in ≥33% of subjects with a DLT

SECONDARY OUTCOMES:
Incidence of Adverse Events [Safety and Tolerability] | Up to Cycle-6 (28-day per cycle)
  Treatment-Emergent Adverse events
Pharmacokinetic (PK) profile of KPG-121 | Cycle-1 (up to 28-day)
  Plasma concentrations of KPG-121

CONTACTS AND LOCATIONS:
Overall Officials: Yao Wang, Study Director — Kangpu Biopharmaceuticals, Ltd.
Locations (3):
- United States (3):
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - North Shore Hematology Oncology Associates DBA NY Cancer and Blood Specialists, Port Jefferson Station, New York
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No